CLINICAL TRIAL: NCT03491397
Title: Safety and Efficacy of Genicular Artery Embolization for the Treatment of Symptomatic Knee Osteoarthritis
Brief Title: Genicular Artery Embolization for the Treatment of Knee Osteoarthritis
Acronym: GAE-OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Siddharth Padia, MD (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor-Investigator, Siddharth Padia, MD, Principal Investigator, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-000560
Record Dates: First submitted 2018-03-23; First posted 2018-04-09 (Actual); Results first posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Knee Osteoarthritis; Degenerative Joint Disease of Knee
Keywords: Microspheres; Artery Embolization; Knee Osteoarthritis; Chronic Pain; Embozene
MeSH Terms: conditions — Osteoarthritis, Knee; Chronic Pain | interventions — Microspheres; Embolization, Therapeutic

STUDY DESIGN:
Intervention Model Description: The stratification will not be randomized, but each category will be limited to 20 patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- GAE OA (Experimental): Subjects will be treated with a genicular artery embolization (GAE) procedure performed with Embozene Microspheres. The microspheres will be delivered in a saline-contrast medium solution and will be delivered to the arteries supplying the areas of the subject's pain.
  Interventions: Device: Embozene MicroSpheres

INTERVENTIONS:
Device: Embozene MicroSpheres — Embozene is a medical device made by Boston Scientific approved in the United States for the treatment of hypervascular tumors and arteriovenous malformations. It consists of thousands of microscopic spheres that are injected into the artery in the knee going to the region of pain. One of the causes of pain in the setting of knee arthritis is increased blood flow going to the specific area of pain. The goal of this procedure is to decrease the blood flow (embolize) to the specific region of the knee that is causing your pain. This is done by infusing Embozene particles into the specific blood vessel (genicular artery) supplying the area of pain in the knee.
  Other Names: Color-Advanced Microspheres; Microspheres for Embolization

SUMMARY:
The purpose of this clinical research study is to examine whether Embozene treatment of the genicular artery is a safe and effective way to treat arthritic knee pain. Embozene is a medical device made by Boston Scientific approved in the United States for the treatment of hypervascular tumors and arteriovenous malformations. It consists of thousands of microscopic spheres that are injected into the artery in the knee going to the region of pain. One of the causes of pain in the setting of knee arthritis is increased blood flow going to the specific area of pain. The goal of this procedure is to decrease the blood flow (embolize) to the specific region of the knee that is causing your pain. This is done by infusing Embozene particles into the specific blood vessel (genicular artery) supplying the area of pain in the knee.

DETAILED DESCRIPTION:
This is a phase 2, single-center, prospective, single arm investigational study to evaluate the safety and efficacy of genicular artery embolization (GAE) for treatment of symptomatic knee osteoarthritis (OA). Subjects will be treated with a genicular artery embolization (GAE) procedure performed with Embozene Microspheres. The microspheres will be delivered in a saline-contrast medium solution and will be delivered to the arteries supplying the areas of the subject's pain. The primary objective of this investigation is to assess safety of genicular artery embolization (GAE) for knee osteoarthritis (OA) using Embozene particles.

ELIGIBILITY:
Inclusion Criteria:

* Provided informed consent
* Age ≥ 40 years and ≤ 80 years
* Life expectancy greater than 12 months
* Ineligibility for or refusal of surgical management
* Moderate-severe knee pain as determined by visual analog scale > 4
* Osteoarthritis based on xray
* Local knee tenderness
* Resistant/failed conservative treatment (e.g. NSAIDS/physical therapy/steroid joint injection)

Exclusion Criteria:• Mild knee pain as determined by visual analog scale < 4

* Chronic renal insufficiency (serum creatinine >2 mg/dL)
* Uncorrectable bleeding diathesis: international normalized ratio (INR) >1.6, Platelets <50,000
* Significant arterial atherosclerosis that would limit selective angiography
* Allergy to iodinated contrast agents that is not responsive to steroid management
* Active Infection or malignancy
* Appropriate candidate for knee replacement surgery determined by clinical and physical examination
* Recent (within 3 months) or active cigarette use

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-02-10 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Siddharth Padia, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- Siddharth Padia, M.D., Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 65 individuals assessed for eligibility, 20 did not meet inclusion criteria and 5 declined to participate
Groups:
- Genicular Artery Embolization (GAE) With Embozene Microspheres: Subjects were treated with a genicular artery embolization (GAE) procedure performed with Embozene Microspheres. The microspheres were delivered in a saline-contrast medium solution and delivered to the arteries supplying the areas of the subject's pain.
Period: Overall Study
Arm/Group | Genicular Artery Embolization (GAE) With Embozene Microspheres
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Genicular Artery Embolization (GAE) With Embozene Microspheres
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 69 [49 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] — Body Mass Index (BMI) is a simple calculation of kg/m^2 where kg is a person's weight in kilograms and m^2 is their height in metres squared. A BMI of 25.0 or more is overweight, while the healthy range is 18.5 to 24.9.
  kg/m^2 | 29.3 [18.8 to 43.7]
WOMAC Index [Median (Full Range); unit: units on a scale] — The The Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index is a self-administered questionnaire consisting of 24 items divided into 3 subscales. Each item is scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). Possible score range 0-96. Higher scores indicate worse pain, stiffness, and functional limitations.
  units on a scale | 52 [23 to 88]
WOMAC Pain Score [Median (Full Range); unit: units on a scale] — The Western Ontario and McMaster Universities Osteoarthritis (WOMAC) pain scale quantifies knee pain severity with activities of daily living. The WOMAC pain scale asks the patient to rate the extent of pain in the involved knee/hip during activities. The WOMAC pain scale ranges from 0 (no pain with all 5 activities, ie, flat surface walking, stairclimbing, at night, sitting or lying, standing) to 20 (extreme pain with all 5 activities).
  units on a scale | 11 [5 to 19]
Visual Analog Scale (VAS) pain score [Median (Full Range); unit: units on a scale] — The severity of knee pain was quantified using a visual analog scale (VAS) score ranging from 0 (indicating no pain) through 10 (indicating the worst pain imaginable).
  units on a scale | 8 [5 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Treatment-related Adverse Events, as a Measure of Safety
Description: Treatment-related AEs from gennicular artery embolization during the study period
Time Frame: Up to 12 Months after GAE
Measure: Count of Participants; unit: Participants
Arm/Group | Genicular Artery Embolization (GAE) With Embozene Microspheres
Number analyzed (Participants) | 40
Participants
  Groin hematoma | 1
  Self-resolving focal skin ulceration | 7
  Asymptomatic small bone infarct on MRI | 2

2. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) as a Measure of Efficacy
Description: The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a self-administered questionnaire consisting of 24 items divided into 3 subscales. Each item is scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). With a total possible range of 0-96, higher scores indicate worse pain, stiffness, and functional limitations.
  Pain (5 items, possible range 0-20): during walking, using stairs, in bed, sitting or lying, and standing upright Stiffness (2 items, possible range 0-8): after first waking and later in the day Physical Function (17 items, possible range 0-68): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties
Time Frame: Baseline, Month 1, Month 3, Month 6, Month 12
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Genicular Artery Embolization (GAE) With Embozene Microspheres
Number analyzed (Participants) | 40
score on a scale
  Month 1 | -20.5 [-71 to 20]
  Month 3 | -29.5 [-74 to 26]
  Month 6 | -26.5 [-81 to 19]
  Month 12 | -29.0 [-82 to 19]

3. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Pain Subscale as a Measure of Efficacy
Description: The WOMAC Pain Subscale is a self-administered questionnaire of 5 items to assess Pain: during walking, using stairs, in bed, sitting or lying, and standing upright.
  Each item is scored on a scale of 0-4: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4), with a possible total score range of 0-20.
Time Frame: Baseline, Month 1, Month 3, Month 6, Month 12
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Genicular Artery Embolization (GAE) With Embozene Microspheres
Number analyzed (Participants) | 40
score on a scale
  Month 1 | -6 [-17 to 3]
  Month 3 | -7 [-15 to 6]
  Month 6 | -7 [-14 to 6]
  Month 12 | -7.5 [-14 to 6]

4. Secondary Outcome: Change From Baseline in Visual Analog Scale (VAS) as a Measure of Efficacy
Description: The patient-reported severity of knee pain was quantified using a visual analog scale (VAS) score ranging from 0 (indicating no pain) through 10 (indicating the worst pain imaginable).
Time Frame: Baseline, Month 1, Month 3, Month 6, Month 12
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Genicular Artery Embolization (GAE) With Embozene Microspheres
Number analyzed (Participants) | 40
score on a scale
  Month 1 | -4.5 [-9 to 2]
  Month 3 | -4.5 [-10 to 2]
  Month 6 | -5.0 [-8.5 to -1]
  Month 12 | -5.0 [-9 to 0]

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse Events were recorded, per protocol, only if determined to be at least possibly related to study intervention
Arm/Group | Genicular Artery Embolization (GAE) With Embozene Microspheres
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 1/40
Other Adverse Events (participants affected / at risk) | 9/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Genicular Artery Embolization (GAE) With Embozene Microspheres (N=40)
Groin hematoma (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Genicular Artery Embolization (GAE) With Embozene Microspheres (N=40)
Focal skin ulceration (Skin and subcutaneous tissue disorders) | 7 (7)
Asymptomatic bone infarct (Musculoskeletal and connective tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-13): https://cdn.clinicaltrials.gov/large-docs/97/NCT03491397/Prot_SAP_000.pdf